CLINICAL TRIAL: NCT06660186
Title: Randomized Trial of Rigid Plate Fixation Versus Wire Cerclage in High-Risk Sternotomy Patients
Brief Title: Sternal Plating High Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20240513
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Heart Diseases
Keywords: Cardiac Surgery; Wound Complication; Rigid Sternal Fixation; Sternal Infection; Pain; Non-union
MeSH Terms: conditions — Heart Diseases; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Rigid Sternal Fixation (Experimental): The surgeon will close the sternum (breastbone) using the SternalPlate system. The SternalPlate System consists of implants and instruments used to hold the two halves of the sternum together.
  Interventions: Device: Rigid Sternal Fixation
- Wire Cerclage (Active Comparator): The surgeon will close the sternum (breastbone) using Wire Cerclage. Wire Cerclage consists of stainless steel wires used to hold the two halves of the sternum together.
  Interventions: Device: Wire Cerclage

INTERVENTIONS:
Device: Rigid Sternal Fixation — The surgeon will close the sternum (breastbone) using the SternalPlate system. The SternalPlate System consists of implants and instruments used to hold the two halves of the sternum together.
  Arms: Rigid Sternal Fixation
Device: Wire Cerclage — The surgeon will close the sternum (breastbone) using Wire Cerclage. Wire Cerclage consists of stainless steel wires used to hold the two halves of your sternum together.
  Arms: Wire Cerclage

SUMMARY:
Participants are being invited to participate in a research study at University Hospitals because they have heart disease and are scheduled for open heart surgery. Currently, UH cardiac surgeons close the sternum (or breastbone) after a sternotomy (procedure that allows a doctor to reach the heart and blood vessels) with either a rigid plate fixation Sternal Plate or a Wire Cerclage. However, the study team would like to further evaluate these two techniques. Any volunteer over the age of 18 who is at an increased risk for developing sternal wound complications may be eligible to participate.

ELIGIBILITY:
Preoperative Inclusion Criteria

* Adults (age range: 18-89)
* Undergoing cardiac surgery through sternotomy

  -≥2 risk factors:
* Diabetes mellitus
* Severe COPD
* Chronic steroid use
* Immunosuppression
* Redo sternotomy
* Chronic
* Kidney disease with GFR >30 ml/min per 1.73m2
* Radiation therapy
* BMI≥35
* High-risk of delirium
* Heavy alcohol use

Preoperative Exclusion Criteria

* Active malignancy
* Chronic narcotic use
* NYHA Class IV
* Known nickel metal allergy
* Compliance concern
* eGFR<30 ml/min per 1.73m2
* Involvement in another interventional clinical trial (non-registry)
* Any criteria precluding RPF or WC

Operative Inclusion Criteria

* Off-midline sternotomy
* BITA grafting
* CPB time ≥120 minutes
* Transverse sternal fracture

Operative Exclusion Criteria

* Emergent or emergent salvage surgery
* Non-standard sternotomies
* Sternotomy with bony margin <2 mm
* Bleeding
* Delayed sternal closure
* Surgical complications
* Any criteria precluding RPF or WC

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Sternal healing as measured by CT scan | 6 months
  5 axial CT slices from a priori-defined anatomic locations are selected by a radiologist. Two additional radiologists then independently score each location using a 6-point scale (0, 1, 2, 3, 4, or 5) with higher scores representing greater healing. Sternal union will be pre-specified as a mean score ≥3 (total score ≥15).
Number of sternal wound complications as measured by patient/physician report | 6 months
  Sternal wound complications will be a composite of wound dehiscence, sternal dehiscence, SSIs, and DSWIs (synonymous with deep SSIs and mediastinitis).
Total index hospitalization cost | 6 months
  Index hospitalization costs (beginning at the time of surgery and ending at initial discharge)
Total cost | 6 months
  All costs after initial discharge through 6 months

SECONDARY OUTCOMES:
Change in pain as measured by the Wong-Baker pain scale | Postoperative days 1, 3, day of discharge (up to 10 days), 1 month, 6 months
  From a scale of 0 (no hurts) to 10 (hurts worst)
Change in prescribed narcotic use as measured by patient report | Postoperative days 1, 3, day of discharge (up to 10 days), 1 month, 6 months
  Evaluating mean morphine equivalent
Change in upper extremity functional index (UEFI) | Discharge (up to 10 days), 1 month, 6 months
  The UEFI is a validated 20 item questionnaire used for quantifying UEF in performing normal daily activities.
Change in quality of life as measured by the EuroQol EQ-5D-5L | Discharge (up to 10 days), 1 month, 6 months
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Number of adverse events as measured by patient report | Up to 6 months
  Adverse events of interest not specified above include: damage to soft tissue, organs, or surrounding structures during closure, need for reoperation, loosening of the wires, screws, or plates, fracture of the wires, screws, or plates, and need for hardware removal (wires, screws, or plates).

CONTACTS AND LOCATIONS:
Overall Officials: Marc Pelletier, MD, Principal Investigator — University Hospitals; Rakesh Arora, MD, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No